CLINICAL TRIAL: NCT00641537
Title: A Phase IIIb, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group, Extension Trial to Evaluate the Safety and Tolerability of Oral Cladribine in Subjects With Relapsing-Remitting Multiple Sclerosis Who Have Completed Trial 25643 (CLARITY)
Brief Title: CLARITY Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27820; 2007-000381-20 (EudraCT Number)
Record Dates: First submitted 2008-03-13; First posted 2008-03-24 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-10

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Cladribine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (8):
- Cladribine Low/Placebo (LLPP) (Placebo Comparator)
  Interventions: Drug: Placebo
- Cladribine High Dose/Placebo (HLPP) (Placebo Comparator)
  Interventions: Drug: Placebo
- Cladribine Low/Low Dose (LLLL) (Experimental)
  Interventions: Drug: Cladribine
- Cladribine High/Low Dose (HLLL) (Experimental)
  Interventions: Drug: Cladribine
- Placebo/Cladribine Low Dose (PPLL) (Experimental)
  Interventions: Drug: Cladribine
- Placebo/No Treatment (No Intervention)
- Cladribine 3.5 mg/kg/No Treatment (No Intervention): Participants who received cladribine 3.5 mg/kg in previous study 25643 (NCT00213135) and completed were enrolled in this extension study and received no cladribine treatment and were followed up for safety assessment for 96 weeks (during the treatment period) and followed up for 24 weeks (during supplemental follow-up period).
- Cladribine 5.25 mg/kg/No Treatment (No Intervention): Participants who received cladribine 5.25 mg/kg in previous study 25643 (NCT00213135) and completed were enrolled in this extension study and received no cladribine treatment and were followed up for safety assessment for 96 weeks (during the treatment period) and followed up for 24 weeks (during supplemental follow-up period).

INTERVENTIONS:
Drug: Cladribine — Participants who received Cladribine 3.5 mg/kg in the previous study 25643 (NCT00213135) and completed will be re-randomized in this extension study and receive cladribine tablet orally as cumulative dose of 0.875 mg/kg over a course of 4 or 5 consecutive days of 28-day period at Week 1, 5, 48, and 52 resulting in total cladribine dose of 3.5 mg/kg during the treatment period of 96 weeks.
  Arms: Cladribine Low/Low Dose (LLLL)
Drug: Placebo — Participants who received Cladribine 3.5 mg/kg in the previous study 25643 (NCT00213135) and completed will be re-randomized in this extension study and receive placebo matched to cladribine tablet 0.875 mg/kg orally administered over a course of 4 or 5 consecutive days of 28-day period at Week 1, 5, 48, and 52 during the treatment period of 96 weeks.
  Arms: Cladribine Low/Placebo (LLPP)
Drug: Cladribine — Participants who received Cladribine 5.25 mg/kg in the previous study 25643 (NCT00213135) and completed will be re-randomized in this extension study and receive cladribine tablet orally as cumulative dose of 0.875 mg/kg over a course of 4 or 5 consecutive days of 28-day period at Week 1, 5, 48, and 52 resulting in total cladribine dose of 3.5 mg/kg during the treatment period of 96 weeks.
  Arms: Cladribine High/Low Dose (HLLL)
Drug: Cladribine — Participants who received placebo in the previous study 25643 (NCT00213135) and completed will be re-randomized in this extension study and receive cladribine tablet orally as cumulative dose of 0.875 mg/kg over a course of 4 or 5 consecutive days of 28-day period at Week 1, 5, 48, and 52 resulting in total cladribine dose of 3.5 mg/kg during the treatment period of 96 weeks.
  Arms: Placebo/Cladribine Low Dose (PPLL)
Drug: Placebo — Participants who received Cladribine 5.25 mg/kg in the previous study 25643 (NCT00213135) and completed will be re-randomized in this extension study and receive placebo matched to cladribine tablet 0.875 mg/kg orally administered over a course of 4 or 5 consecutive days of 28-day period at Week 1, 5, 48, and 52 during the treatment period of 96 weeks.
  Arms: Cladribine High Dose/Placebo (HLPP)

SUMMARY:
The purpose of this extension trial was to further evaluate the safety and tolerability of oral cladribine in subjects who have previously completed treatment within Trial 25643 (CLARITY). This trial also explored clinical benefit of prolonged 192-week versus 96-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Randomized in Trial 25643 and satisfied one of the following:

  * Completed randomized treatment course and scheduled visits for the full 96 weeks; or
  * Did not complete the randomized treatment course in Trial 25643 but elected to receive rescue treatment with Rebif®, another beta-interferon, or glatiramer acetate and completed scheduled clinic visits for the full 96 weeks; or
  * Did not complete the randomized treatment course in Trial 25643, declined rescue with Rebif®, another beta-interferon, or glatiramer acetate and still completed scheduled clinic visits for the full 96 weeks; or
  * Did not complete the randomized treatment course in Trial 25643, were not eligible for rescue option with Rebif®, and still completed scheduled clinic visits for the full 96 weeks
* Male or female, between 18 and 65 years of age (inclusive, at time of informed consent for Trial 25643)
* No medical history or evidence of latent tuberculosis infection (LTBI) or tuberculosis (TB), as evidenced by TB skin test or chest X-ray
* All of the following laboratory hematologic parameters evaluated as normal (as define below, inclusively) within 28 days of first dosing of blinded study medication at study Day 1:

  * Hemoglobin = 11.6 to 16.2 gram per deciliter (g/dL)
  * Leukocytes (total white blood cell) = 4.1 to 12.3*10^3 per microliter
  * Absolute lymphocyte count (ALC) = 1.02 to 3.36*10^3 per microliter
  * Absolute neutrophil count (ANC) = 2.03 to 8.36*10^3 per microliter
  * Platelet count = 140 to 450*10^3 per microliter
* Other protocol-defined inclusion/exclusion criteria may apply

Exclusion Criteria:

* Participants who were not enrolled in Trial 25643
* Participant has moderate to severe renal impairment
* Use of mitoxantrone, total lymphoid irradiation, myelosuppressive therapy, campath-1h, cyclophosphamide, azathioprine, methotrexate or natalizumab at any time during and since Trial 25643
* Use of cytokine or anti-cytokine therapy, intravenous immunoglobulin (IVIG) or plasmapheresis at any time during and since Trial 25643
* Treatment with oral or systemic corticosteroids or adrenocorticotropic hormone within 28 days before Study Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 867 (Actual)
Dates: Start 2008-02-29 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (116):
- United States (17):
  - Research Site, Boulder, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Northbrook, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Henderson, Nevada
  - Research Site, Newark, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Charleston, West Virginia
- Australia (3):
  - Research Site, Camperdown
  - Research Site, Melbourne
  - Research Site, Victoria
- Research Site, Linz, Austria
- Belgium (2):
  - Research Site, Diepenbeek
  - Research Site, Esneux
- Research Site, Recife, Brazil
- Bulgaria (7):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Shuman
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Zagora
- Canada (4):
  - Research Site, Burnaby
  - Research Site, Greenfield Park
  - Research Site, Ottawa
  - Research Site, Québec
- Croatia (3):
  - Research Site, Karlovac
  - Research Site, Sisak
  - Research Site, Split
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- Research Site, Copenhagen, Denmark
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (2):
  - Research Site, Oulu
  - Research Site, Turku
- France (7):
  - Research Site, Clermont-Ferrand
  - Research Site, Lille
  - Research Site, Nancy
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Saint-Herblain
- Germany (6):
  - Research Site, Bochum
  - Research Site, Frankfurt
  - Research Site, Giessen
  - Research Site, Hanover
  - Research Site, Regensburg
  - Research Site, Rostock
- Research Site, Athens, Greece
- Italy (9):
  - Research Site, Bari
  - Research Site, Cagliari
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
- Research Site, Riga, Latvia
- Research Site, Beirut, Lebanon
- Research Site, Kaunas, Lithuania
- Morocco (3):
  - Research Site, Casablanca
  - Research Site, Fes
  - Research Site, Rabat
- Research Site, Sittard- Geleen, Netherlands
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warszawy
- Research Site, Lisbon, Portugal
- Russia (15):
  - Research Site, Kaluga
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Reseach Site, Saratov
  - Research Site, Tomsk
  - Research Site, Vladimir
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Research Site, Riyadh, Saudi Arabia
- Research Site, Belgrade, Serbia
- Switzerland (2):
  - Research Site, Lausanne
  - Research Site, Sankt Gallen
- Tunisia (3):
  - Research Site, Monastir
  - Research Site, Sfax
  - Research Site, Tunis
- Turkey (Türkiye) (2):
  - Research Site, Bursa
  - Research Site, Izmir
- Ukraine (4):
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Lviv
  - Research Site, Vinnitsa
- United Kingdom (6):
  - Research Site, Hull
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Sheffield
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Derived] Stefano N, Sormani MP, Giovannoni G, Rammohan K, Leist TP, Coyle PK, Dangond F, Alexandri N, Galazka A. Relapses in people with multiple sclerosis treated with cladribine tablets followed for up to 5 years: a plain language summary. Neurodegener Dis Manag. 2022 Dec;12(6):303-310. doi: 10.2217/nmt-2022-0019. Epub 2022 Aug 26. PMID 36017797
- [Derived] Giovannoni G, Comi G, Rammohan K, Rieckmann P, Dangond F, Jack D, Vermersch P. Disease stability over five years in people with multiple sclerosis treated with cladribine tablets: a plain language summary. Neurodegener Dis Manag. 2022 Dec;12(6):295-301. doi: 10.2217/nmt-2022-0018. Epub 2022 Aug 26. PMID 36017780
- [Derived] Giovannoni G, Coyle PK, Vermersch P, Walker B, Aldridge J, Nolting A, Galazka A, Lemieux C, Leist TP. Integrated Lymphopenia Analysis in Younger and Older Patients With Multiple Sclerosis Treated With Cladribine Tablets. Front Immunol. 2021 Dec 24;12:763433. doi: 10.3389/fimmu.2021.763433. eCollection 2021. PMID 35003076
- [Derived] Giovannoni G, Comi G, Rammohan K, Rieckmann P, Dangond F, Keller B, Jack D, Vermersch P. Long-Term Disease Stability Assessed by the Expanded Disability Status Scale in Patients Treated with Cladribine Tablets 3.5 mg/kg for Relapsing Multiple Sclerosis: An Exploratory Post Hoc Analysis of the CLARITY and CLARITY Extension Studies. Adv Ther. 2021 Sep;38(9):4975-4985. doi: 10.1007/s12325-021-01865-w. Epub 2021 Aug 9. PMID 34370275
- [Derived] De Stefano N, Sormani MP, Giovannoni G, Rammohan K, Leist T, Coyle PK, Dangond F, Keller B, Alexandri N, Galazka A. Analysis of frequency and severity of relapses in multiple sclerosis patients treated with cladribine tablets or placebo: The CLARITY and CLARITY Extension studies. Mult Scler. 2022 Jan;28(1):111-120. doi: 10.1177/13524585211010294. Epub 2021 May 10. PMID 33969750
- [Derived] Giovannoni G, Galazka A, Schick R, Leist T, Comi G, Montalban X, Damian D, Dangond F, Cook S. Pregnancy Outcomes During the Clinical Development Program of Cladribine in Multiple Sclerosis: An Integrated Analysis of Safety. Drug Saf. 2020 Jul;43(7):635-643. doi: 10.1007/s40264-020-00948-x. PMID 32447743
- [Derived] Comi G, Cook S, Rammohan K, Soelberg Sorensen P, Vermersch P, Adeniji AK, Dangond F, Giovannoni G. Long-term effects of cladribine tablets on MRI activity outcomes in patients with relapsing-remitting multiple sclerosis: the CLARITY Extension study. Ther Adv Neurol Disord. 2018 Jan 23;11:1756285617753365. doi: 10.1177/1756285617753365. eCollection 2018. PMID 29399054
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=27820
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1326 subjects were randomized into CLARITY from study 25643 (NCT00213135), of whom 867 consented to participate in this phase 3b extension Study 27820. 806 subjects were randomized or assigned to treatment and a further 61 subjects were followed for safety only (Supplemental follow-up period [no study treatment] [SAFUP]).
Groups:
- Cladribine Low/Placebo (LLPP): Participants who received cladribine 3.5 mg/kg in previous study 25643 (NCT00213135) and completed the study who were randomized or assigned to placebo (matched to cladribine tablet) during the treatment period of 96 weeks. Participants were followed up for 24 weeks in Supplemental follow-up period (SUPF).
- Cladribine High Dose/Placebo (HLPP): Participants who received cladribine 5.25 mg/kg in previous study 25643 (NCT00213135) and completed the study who were randomized or assigned to placebo (matched to cladribine tablet) during the treatment period of 96 weeks. Participants were followed up for 24 weeks in SUPF.
- Cladribine Low/Low Dose (LLLL): Participants who received cladribine 3.5 mg/kg in previous study 25643 (NCT00213135) and completed the study who were randomized or assigned to cladribine 3.5 mg/kg orally provided as 0.875 mg/kg treatment weeks at Week 1, Week 5, Week 48 and Week 52 resulting in total dose of 3.5 mg/kg during the treatment period of 96 weeks. Participants were followed up for 24 weeks in SUPF.
- Cladribine High/Low Dose (HLLL): Participants who received cladribine 5.25 mg/kg in previous study 25643 (NCT00213135) and completed the study who were randomized or assigned to cladribine 3.5 mg/kg orally provided as 0.875 mg/kg treatment weeks at Week 1, Week 5, Week 48 and Week 52 resulting in total dose of 3.5 mg/kg during the treatment period of 96 weeks. Participants were followed up for 24 weeks in SUPF.
- Placebo/Cladribine Low Dose (PPLL): Participants who received placebo in previous study 25643 (NCT00213135) and completed the study who were randomized or assigned to cladribine 3.5 mg/kg orally provided as 0.875 mg/kg treatment weeks at Week 1, Week 5, Week 48 and Week 52 resulting in total dose of 3.5 mg/kg during the treatment period of 96 weeks. Participants were followed up for 24 weeks in SUPF.
- Placebo/No Treatment: Participants who received placebo matched to cladribine in previous study 25643 (NCT00213135) and were enrolled in this extension study and received no cladribine treatment and were followed up for safety assessment for 96 weeks (during the treatment period) and followed up for 24 weeks (during supplemental follow-up period).
Period: 96-week Period
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL) | Placebo/No Treatment | Cladribine 3.5 mg/kg/No Treatment | Cladribine 5.25 mg/kg/No Treatment
Started | 98 | 92 | 186 | 186 | 244 | 22 | 17 | 22
Completed | 89 | 82 | 166 | 174 | 227 | 15 | 12 | 16
Not Completed | 9 | 10 | 20 | 12 | 17 | 7 | 5 | 6
Not completed — Adverse Event | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 2 | 2 | 4 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Death | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 7 | 14 | 9 | 11 | 6 | 4 | 6
Period: 24-Week Supplemental Follow-up Period
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL) | Placebo/No Treatment | Cladribine 3.5 mg/kg/No Treatment | Cladribine 5.25 mg/kg/No Treatment
Started | 75 | 69 | 143 | 151 | 198 | 15 | 9 | 11
Completed | 75 | 66 | 140 | 147 | 193 | 14 | 8 | 10
Not Completed | 0 | 3 | 3 | 4 | 5 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 3 | 2 | 1 | 0 | 0
Not completed — Other | 0 | 2 | 2 | 1 | 3 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL) | Total
Number analyzed (Participants) | 98 | 92 | 186 | 186 | 244 | 806
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (10.7) | 40.8 (9.6) | 40.6 (10.5) | 41.4 (10.1) | 41.6 (9.6) | 41.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 59 | 124 | 125 | 156 | 531
  Male | 31 | 33 | 62 | 61 | 88 | 275

OUTCOME MEASURES:

1. Primary Outcome: Safety Population: Percentage of Participants With at Least 1 Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE) Grade 4 Hematologic and Hepatic Toxicity
Description: Hematologic and hepatic toxicity was assessed using Common Terminology Criteria for Adverse Events v 3.0 (CTCAE). Hematologic and hepatic function included absolute lymphocyte count (ALC), hemoglobin level, white blood cell (WBC) count, absolute neutrophil count (ANC), platelets, alanine transaminase (ALT), aspartate transaminase (AST) and bilirubin. According to CTCAE v3.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death.
Time Frame: Baseline up to Week 120
Population: Safety population included all the randomized participants who had received at least 1 dose of study medication and had follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 98 | 92 | 186 | 186 | 244
percentage of participants
  Lymphocyte toxicity | 0.0 | 0.0 | 2.7 | 3.2 | 0.4
  Hemoglobin Toxicity | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  White Blood Cell Toxicity | 0.0 | 0.0 | 0.5 | 0.0 | 0.0
  Absolute Neutrophil Count Toxicity | 0.0 | 2.2 | 0.5 | 0.0 | 0.4
  Platelets Toxicity | 0.0 | 0.0 | 0.5 | 0.0 | 0.0
  Alanine Transaminase Toxicity | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  AsparateTransaminase Toxicity | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Bilirubin Toxicity | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

2. Primary Outcome: Safety Population: Mean Change From Baseline in Absolute Lymphocyte Count, Platelet, Neutrophils and Leukocytes at Week 120
Description: Mean change from baseline in absolute lymphocyte count, platelet, neutrophils and leukocytes at week 120 were reported.
Time Frame: Baseline, Week 120
Population: Safety population included all the randomized participants who had received at least 1 dose of study medication and had follow-up safety data. Here 'Number of participants analyzed' signifies number of participants who were evaluable for this outcome measure and "Number analyzed" are those who were evaluable at specified category.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 73 | 62 | 137 | 144 | 187
10^9 cells per liter
  Lymphocyte Count: number analyzed (Participants) | 73 | 62 | 137 | 142 | 187
  Lymphocyte Count | 0.3 (0.4) | 0.3 (0.4) | 0.0 (0.4) | 0.0 (0.5) | -0.6 (0.6)
  Platelet: number analyzed (Participants) | 73 | 62 | 136 | 143 | 187
  Platelet | -7.7 (26.2) | -11.9 (35.3) | -20.6 (37.9) | -9.7 (51.2) | -34.0 (37.2)
  Leukocytes: number analyzed (Participants) | 73 | 62 | 136 | 144 | 187
  Leukocytes | 0.8 (1.5) | 0.5 (1.2) | -0.2 (1.5) | -0.1 (1.4) | -0.9 (1.7)
  Neutrophils: number analyzed (Participants) | 73 | 62 | 137 | 142 | 187
  Neutrophils | 0.4 (1.3) | 0.1 (1.2) | -0.2 (1.4) | -0.2 (1.3) | -0.3 (1.7)

3. Primary Outcome: Safety Population: Mean Change From Baseline in Hemoglobin at Week 120
Description: Mean change from baseline in hemoglobin at Week 120 was reported.
Time Frame: Baseline, Week 120
Population: Safety population included all the randomized participants who had received at least 1 dose of study medication and had follow-up safety data. Here 'Number of participants analyzed' signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 73 | 62 | 137 | 144 | 187
grams per deciliter (g/dL) | 0.2 (0.9) | 0.2 (0.7) | -0.1 (0.9) | 0.1 (0.9) | -0.1 (0.9)

4. Primary Outcome: Safety Population: Mean Change From Baseline in Aspartate Aminotransferase and Alanine Aminotransferase at Week 120
Description: Mean change from baseline in aspartate aminotransferase and alanine aminotransferase at week 120 were reported.
Time Frame: Baseline, Week 120
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units per litre (U/L)
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 72 | 62 | 137 | 142 | 185
Units per litre (U/L)
  Aspartate Aminotransferase: number analyzed (Participants) | 72 | 62 | 137 | 142 | 184
  Aspartate Aminotransferase | 0.7 (10.6) | -1.1 (6.4) | 2.2 (7.3) | 0.7 (11.3) | 0.5 (5.1)
  Alanine Aminotransferase | 2.2 (26.0) | -1.0 (11.7) | 4.3 (14.3) | 0.7 (17.5) | 1.4 (12.2)

5. Primary Outcome: Safety Population: Mean Change From Baseline in Bilirubin at Week 120
Description: Mean Change From Baseline in Bilirubin at week 120 was reported.
Time Frame: Baseline, Week 120
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micromoles per liter (mcmol/L)
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 73 | 62 | 137 | 144 | 186
micromoles per liter (mcmol/L) | 0.1 (3.7) | 0.0 (3.5) | -0.8 (3.7) | -0.8 (3.3) | -0.4 (3.7)

6. Primary Outcome: Safety Population: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered. Serious AE (SAE): Any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. Number of participants with TEAEs included participants with both non-serious TEAEs and serious TEAEs.
Time Frame: Baseline up to Week 120
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 98 | 92 | 186 | 186 | 244
Participants
  TEAEs | 74 | 71 | 149 | 149 | 194
  Serious TEAEs | 16 | 8 | 25 | 23 | 22

7. Primary Outcome: SAFUP Analysis Set: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered. SAE: Any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. Number of participants with TEAEs included participants with both non-serious TEAEs and serious TEAEs.
Time Frame: Baseline up to Week 120
Population: SAFUP Analysis Set included all participants who were enrolled and had at least one safety assessment, but were not randomized or assigned to treatment because they were not eligible to receive study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/No Treatment | Cladribine 3.5 mg/kg/No Treatment | Cladribine 5.25 mg/kg/No Treatment
Number analyzed (Participants) | 22 | 17 | 22
Participants
  TEAEs | 16 | 13 | 18
  Serious TEAEs | 2 | 1 | 3

8. Primary Outcome: Safety Population: Number of Participants Who Developed Infections (Herpes Viral Infection, Viral Infectious Disorder and Opportunistic Infection), Infection-related Adverse Events and Malignancies
Description: Number of participants who developed Herpes viral infection, Viral infectious disorder and Opportunistic infection are reported. Number of participants with infection related adverse events are the number of participants who had at least one adverse event coded to medical dictionary for regulatory activities (MedDRA) preferred terms under infection and infestation system organ class. Malignancy is defined as having at least one adverse event coded to MedDRA preferred terms under the pre-specified grouping Malignant and unspecified tumors.
Time Frame: Baseline up to Week 120
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 98 | 92 | 186 | 186 | 244
Participants
  Herpes viral infection | 6 | 4 | 6 | 13 | 11
  Opportunistic infection | 8 | 4 | 9 | 17 | 15
  Viral infectious disorder | 20 | 16 | 28 | 41 | 39
  Infections related adverse event | 49 | 45 | 92 | 88 | 112
  Malignancies | 2 | 1 | 7 | 2 | 2

9. Primary Outcome: SAFUP Analysis Set: Number of Participants Who Developed Infections (Herpes Viral Infection, Viral Infectious Disorder and Opportunistic Infection), Infection-related Adverse Events and Malignancies
Description: Number of participants who developed Herpes viral infection, Viral infectious disorder and Opportunistic infection were reported. Number of participants with infection related adverse events are the number of participants who had at least one adverse event coded to medical dictionary for regulatory activities (MedDRA) preferred terms under infection and infestation system organ class. Malignancy is defined as having at least one adverse event coded to MedDRA preferred terms under the pre-specified grouping Malignant and unspecified tumors.
Time Frame: Baseline up to Week 120
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/No Treatment | Cladribine 3.5 mg/kg/No Treatment | Cladribine 5.25 mg/kg/No Treatment
Number analyzed (Participants) | 22 | 17 | 22
Participants
  Herpes viral infection | 0 | 1 | 1
  Opportunistic infection | 0 | 1 | 2
  Viral infectious disorder | 6 | 5 | 3
  Infections related adverse event | 11 | 6 | 12
  Malignancies | 2 | 0 | 1

10. Primary Outcome: Safety Population: Time to First Grade 3 or 4 Hematological Toxicity and Liver Toxicity
Description: Hematologic and hepatic toxicity was assessed using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE). Hematologic and hepatic function included absolute lymphocyte count (ALC), hemoglobin level, white blood cell (WBC) count, absolute neutrophil count (ANC), platelets, alanine transaminase (ALT), aspartate transaminase (AST) and bilirubin. Time to first CTCAE Grade 3 or 4 hematological or liver toxicity was analyzed by treatment group using Kaplan-Meier plots of probability of surviving toxicity-free and point estimates of percentiles. According to CTCAE version 3.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death. 10th, 20th, 25th, 50th and 75th percentiles were estimated from Kaplan-Meier survival curve.
Time Frame: Baseline up to Week 120
Population: Safety population included all the randomized participants who had received at least 1dose of study medication and had follow-up safety data. Here 'Number of participants analyzed' signifies number of participants who were evaluable for this outcome measure and "Number Analyzed"signifies those participants who were evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 5 | 6 | 76 | 99 | 61
Days
  10th percentile: Lymphocytes Count | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | 14 [8 to 34] | 8 [8 to 12] | 362 [85 to 378]
  20th percentile: Lymphocytes Count | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | 58 [34 to 162] | 15 [12 to 50] | 412 [379 to 583]
  25th percentile: Lymphocytes Count | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | 108 [57 to 379] | 34 [15 to 57] | 583 [406 to NA] — Due to higher percentiles not attained, upper limit of 95% Confidence Interval from the Kaplan-Meier survival curves could not be derived.
  50th percentile: Lymphocytes Count | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | 449 [361 to NA] — Due to higher percentiles not attained, upper limit of 95% Confidence Interval from the Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  75th percentile: Lymphocytes Count | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: Hemoglobin: number analyzed (Participants) | 0 | 1 | 2 | 1 | 3
  10th percentile: Hemoglobin |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: Hemoglobin: number analyzed (Participants) | 0 | 1 | 2 | 1 | 3
  20th percentile: Hemoglobin |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  25th percentile: Hemoglobin: number analyzed (Participants) | 0 | 1 | 2 | 1 | 3
  25th percentile: Hemoglobin |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  50th percentile: Hemoglobin: number analyzed (Participants) | 0 | 1 | 2 | 1 | 3
  50th percentile: Hemoglobin |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  75th percentile: Hemoglobin: number analyzed (Participants) | 0 | 1 | 2 | 1 | 3
  75th percentile: Hemoglobin |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: WBC: number analyzed (Participants) | 0 | 1 | 11 | 11 | 5
  10th percentile: WBC |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: WBC: number analyzed (Participants) | 0 | 1 | 11 | 11 | 5
  20th percentile: WBC |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  25th percentile: WBC: number analyzed (Participants) | 0 | 1 | 11 | 11 | 5
  25th percentile: WBC |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  50th percentile: WBC: number analyzed (Participants) | 0 | 1 | 11 | 11 | 5
  50th percentile: WBC |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  75th percentile: WBC: number analyzed (Participants) | 0 | 1 | 11 | 11 | 5
  75th percentile: WBC |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: ANC: number analyzed (Participants) | 4 | 3 | 11 | 12 | 8
  10th percentile: ANC | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: ANC: number analyzed (Participants) | 4 | 3 | 11 | 12 | 8
  20th percentile: ANC | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  25th percentile: ANC: number analyzed (Participants) | 4 | 3 | 11 | 12 | 8
  25th percentile: ANC | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  50th percentile: ANC: number analyzed (Participants) | 4 | 3 | 11 | 12 | 8
  50th percentile: ANC | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  75th percentile: ANC: number analyzed (Participants) | 4 | 3 | 11 | 12 | 8
  75th percentile: ANC | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: Platelets: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  10th percentile: Platelets |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  20th percentile: Platelets: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  20th percentile: Platelets |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  25th percentile: Platelets: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  25th percentile: Platelets |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  50th percentile: Platelets: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  50th percentile: Platelets |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  75th percentile: Platelets: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  75th percentile: Platelets |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |
  10th percentile: ALT: number analyzed (Participants) | 2 | 0 | 0 | 3 | 3
  10th percentile: ALT | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: ALT: number analyzed (Participants) | 2 | 0 | 0 | 3 | 3
  20th percentile: ALT | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  25th percentile: ALT: number analyzed (Participants) | 2 | 0 | 0 | 3 | 3
  25th percentile: ALT | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  50th percentile: ALT: number analyzed (Participants) | 2 | 0 | 0 | 3 | 3
  50th percentile: ALT | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  75th percentile: ALT: number analyzed (Participants) | 2 | 0 | 0 | 3 | 3
  75th percentile: ALT | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: AST: number analyzed (Participants) | 2 | 0 | 1 | 1 | 1
  10th percentile: AST | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  20th percentile: AST: number analyzed (Participants) | 2 | 0 | 1 | 1 | 1
  20th percentile: AST | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  25th percentile: AST: number analyzed (Participants) | 2 | 0 | 1 | 1 | 1
  25th percentile: AST | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  50th percentile: AST: number analyzed (Participants) | 2 | 0 | 1 | 1 | 1
  50th percentile: AST | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  75th percentile: AST: number analyzed (Participants) | 2 | 0 | 1 | 1 | 1
  75th percentile: AST | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. |  | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived. | NA [NA to NA] — Due to small number of events, estimates from Kaplan-Meier survival curves could not be derived.
  10th percentile: Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  20th percentile: Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  25th percentile: Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  50th percentile: Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  75th percentile: Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Safety Population: Median Time to Recovery From Grade 3 or 4 Hematological and Hepatic Toxicity
Description: Hematologic and hepatic toxicity was assessed using Common Terminology Criteria for Adverse Events (CTCAE). Hematologic and hepatic function included absolute lymphocyte count (ALC), hemoglobin level, white blood cell (WBC) count, absolute neutrophil count (ANC), platelets, alanine transaminase (ALT), aspartate transaminase (AST) and bilirubin. According to CTCAE version 3.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death. Time to recovery from grade 3 or 4 hematological or liver toxicity were reported: lymphocytes, platelets, neutrophils, white blood cells, hemoglobin, Alanine transaminase (ALT), Aspartate transaminase (AST), Platelets and Bilirubin. Recovery from a Grade 3 or 4 toxicity is defined as a return to a Grade 0 or 1.
Time Frame: Baseline up to Week 120
Population: Safety population included all the randomized participants who had received at least 1dose of study medication and had follow-up safety data. Here 'Number of participants analyzed' signifies number of participants who were evaluable for this outcome measure and "Number Analyzed signifies those participants who were evaluable for specified category.
Measure: Median (Full Range); unit: Days
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 5 | 4 | 69 | 89 | 50
Days
  Lymphocyte | 22.0 [14 to 85] | 31.5 [26 to 51] | 212.0 [8 to 1184] | 168.0 [7 to 799] | 111.3 [5 to 701]
  Hemoglobin: number analyzed (Participants) | 0 | 1 | 1 | 1 | 2
  Hemoglobin |  | 99.0 [99 to 99] | 64.0 [64 to 64] | 57.0 [57 to 57] | 173.5 [22 to 325]
  White Blood Cell Count: number analyzed (Participants) | 0 | 1 | 9 | 10 | 5
  White Blood Cell Count |  | 29.0 [29 to 29] | 30.0 [19 to 295] | 42.5 [19 to 715] | 79.0 [28 to 125]
  Absolute Neutrophil Count: number analyzed (Participants) | 3 | 2 | 6 | 11 | 6
  Absolute Neutrophil Count | 43.0 [13 to 91] | 57.0 [29 to 85] | 23.8 [8 to 85] | 34.0 [19 to 127] | 37.5 [15 to 162]
  Platelets: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Platelets |  |  |  | 197.0 [197 to 197] |
  Alanine Transaminase (ALT): number analyzed (Participants) | 2 | 0 | 0 | 2 | 3
  Alanine Transaminase (ALT) | 72.5 [51 to 94] |  |  | 73.0 [19 to 127] | 15.0 [1 to 55]
  Aspartate Transaminase (AST): number analyzed (Participants) | 2 | 0 | 1 | 1 | 1
  Aspartate Transaminase (AST) | 72.5 [51 to 94] |  | 84.0 [84 to 84] | 18.0 [18 to 18] | 55.0 [55 to 55]
  Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Safety Population: Mean Time to Recovery From Grade 3 or 4 Hematological and Liver Toxicity
Description: Hematologic and hepatic toxicity was assessed using Common Terminology Criteria for Adverse Events (CTCAE). Hematologic and hepatic function included absolute lymphocyte count (ALC), hemoglobin level, white blood cell (WBC) count, absolute neutrophil count (ANC), platelets, alanine transaminase (ALT), aspartate transaminase (AST) and bilirubin. According to CTCAE v3.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death. Time to recovery from grade 3 or 4 hematological or liver toxicity were reported: lymphocytes, platelets, neutrophils, white blood cells, hemoglobin, Alanine transaminase (ALT), Aspartate transaminase (AST) and Platelets. Recovery from a Grade 3 or 4 toxicity is defined as a return to a Grade 0 or 1.
Time Frame: Baseline up to Week 120
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 5 | 4 | 69 | 89 | 50
Days
  Lymphocyte | 41.0 (33.5) | 34.9 (11.7) | 256.7 (239.7) | 241.8 (216.1) | 160.2 (160.4)
  Hemoglobin: number analyzed (Participants) | 0 | 1 | 1 | 1 | 2
  Hemoglobin |  | 99.0 | 64.0 | 57.0 | 173.5 (214.3)
  White Blood Cell Count: number analyzed (Participants) | 0 | 1 | 9 | 10 | 5
  White Blood Cell Count |  | 29.0 | 79.3 (91.9) | 132.0 (213.9) | 71.5 (39.7)
  Absolute Neutrophil Count: number analyzed (Participants) | 3 | 2 | 6 | 11 | 6
  Absolute Neutrophil Count | 49.0 (39.3) | 57.0 (39.6) | 35.3 (29.9) | 46.8 (35.1) | 61.0 (55.3)
  Platelets: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Platelets |  |  |  | 197.0 |
  Alanine Transaminase: number analyzed (Participants) | 2 | 0 | 0 | 2 | 3
  Alanine Transaminase | 72.5 (30.4) |  |  | 73.0 (76.4) | 23.7 (28.0)
  Aspartate Transaminase: number analyzed (Participants) | 2 | 0 | 1 | 1 | 1
  Aspartate Transaminase | 72.5 (30.4) |  | 84.0 | 18.0 | 55.0
  Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Safety Population: Median Time to Nadir of Absolute Lymphocyte Count
Description: Median time to nadir of absolute lymphocyte count was reported.
Time Frame: Baseline up to Week 120
Population: as for outcome 3
Measure: Median (97.5% Confidence Interval); unit: Days
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 54 | 57 | 177 | 175 | 227
Days | 162.0 [86 to 372] | 93.0 [37 to 252] | 365.0 [246 to 379] | 162.0 [106 to 359] | 380.0 [379 to 400]

14. Primary Outcome: Safety Population: Mean Time to Nadir of Absolute Lymphocyte Count
Description: Mean time to nadir of absolute lymphocyte count was reported.
Time Frame: Baseline up to Week 120
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 54 | 57 | 177 | 175 | 227
Days | 292.0 (296.7) | 193.6 (219.1) | 276.7 (191.7) | 241.1 (200.3) | 362.9 (177.5)

15. Primary Outcome: Safety Population: Mean Time to Recovery From Nadir of Absolute Lymphocyte Count to Normal Value
Description: Mean time to recovery from nadir of absolute lymphocyte count to normal was reported. Recovery from Nadir is defined as a return to baseline value. Normal absolute lymphocyte count is 1.02 x 10^3 cells/microliter.
Time Frame: Baseline up to Week 120
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 47 | 52 | 130 | 128 | 185
Days | 79.0 (72.4) | 72.7 (61.3) | 237.5 (214.7) | 245.3 (222.3) | 187.8 (180.9)

16. Primary Outcome: Safety Population: Mean Change in Corrected QT (QTc) Interval From Baseline
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. Mean change in corrected QT (QTc) interval from baseline was reported.
Time Frame: Baseline, Week 5, 48, 52 and 96
Population: Safety population included all the randomized participants who had received at least 1 dose of study medication and had follow-up safety data. Here 'Number of participants analyzed' signifies number of participants who were evaluable for this outcome measure and and "Number analyzed" are those who were evaluable at specified category.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL)
Number analyzed (Participants) | 25 | 18 | 31 | 35 | 41
milliseconds
  Week 5 | 7.0 (21.6) | 7.4 (21.2) | 4.5 (20.6) | 4.3 (16.2) | 0.7 (18.8)
  Week 48: number analyzed (Participants) | 19 | 15 | 23 | 33 | 36
  Week 48 | 16.9 (18.6) | 7.4 (23.6) | 9.3 (19.8) | 11.3 (19.5) | 7.2 (19.6)
  Week 52: number analyzed (Participants) | 7 | 3 | 7 | 10 | 11
  Week 52 | 14.9 (17.5) | 22.3 (25.4) | 8.4 (22.8) | 5.2 (18.8) | -1.2 (16.6)
  Week 96: number analyzed (Participants) | 19 | 9 | 24 | 31 | 32
  Week 96 | 5.8 (25.5) | -4.5 (32.5) | -12.5 (22.2) | 1.6 (22.7) | -6.2 (19.2)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 120
Description: For LLPP, HLPP, LLLL, HLLL and PPLL arms: Safety population included all the randomized participants who had received at least 1dose of study medication and had follow-up safety data. For Placebo/No treatment, Cladribine 3.5 mg/kg/No Treatment and Cladribine 5.25 mg/kg/No Treatment: SAFUP Analysis Set included all participants who were enrolled and had at least one safety assessment, but were not randomized or assigned to treatment because they were not eligible to receive study medication.
Arm/Group | Cladribine Low/Placebo (LLPP) | Cladribine High Dose/Placebo (HLPP) | Cladribine Low/Low Dose (LLLL) | Cladribine High/Low Dose (HLLL) | Placebo/Cladribine Low Dose (PPLL) | Placebo/No Treatment | Cladribine 3.5 mg/kg/No Treatment | Cladribine 5.25 mg/kg/No Treatment
All-Cause Mortality (participants affected / at risk) | 2/98 | 0/92 | 1/186 | 0/186 | 0/244 | 0/22 | 0/17 | 0/22
Serious Adverse Events (participants affected / at risk) | 16/98 | 8/92 | 25/186 | 23/186 | 22/244 | 2/22 | 1/17 | 3/22
Other Adverse Events (participants affected / at risk) | 73/98 | 69/92 | 143/186 | 146/186 | 192/244 | 16/22 | 13/17 | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine Low/Placebo (LLPP) (N=98) | Cladribine High Dose/Placebo (HLPP) (N=92) | Cladribine Low/Low Dose (LLLL) (N=186) | Cladribine High/Low Dose (HLLL) (N=186) | Placebo/Cladribine Low Dose (PPLL) (N=244) | Placebo/No Treatment (N=22) | Cladribine 3.5 mg/kg/No Treatment (N=17) | Cladribine 5.25 mg/kg/No Treatment (N=22)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urethral abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drowning (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood culture positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tuberculin test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Secondary immunodeficiency (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venous Stasis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cladribine Low/Placebo (LLPP) (N=98) | Cladribine High Dose/Placebo (HLPP) (N=92) | Cladribine Low/Low Dose (LLLL) (N=186) | Cladribine High/Low Dose (HLLL) (N=186) | Placebo/Cladribine Low Dose (PPLL) (N=244) | Placebo/No Treatment (N=22) | Cladribine 3.5 mg/kg/No Treatment (N=17) | Cladribine 5.25 mg/kg/No Treatment (N=22)
Lymphopenia (Blood and lymphatic system disorders) | 9 | 7 | 68 | 75 | 69 | 2 | 2 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 19 | 20 | 12 | 2 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 7 | 10 | 7 | 1 | 1/5 | 5
Vertigo (Ear and labyrinth disorders) | 5 | 1 | 6 | 5 | 5 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 6 | 9 | 14 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 4 | 11 | 7 | 10 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 4 | 6 | 5 | 3 | 4 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 5 | 5 | 0 | 4 | 0 | 0 | 1
Fatigue (General disorders) | 5 | 5 | 8 | 10 | 12 | 1 | 2 | 1
Influenza like illness (General disorders) | 5 | 2 | 14 | 9 | 10 | 1 | 2 | 2
Nasopharyngitis (Infections and infestations) | 19 | 15 | 22 | 28 | 45 | 1 | 0 | 6
Influenza (Infections and infestations) | 11 | 10 | 15 | 23 | 17 | 4 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 9 | 17 | 20 | 19 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 6 | 4 | 17 | 16 | 16 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 9 | 16 | 18 | 28 | 1 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 6 | 10 | 10 | 11 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 5 | 8 | 13 | 0 | 1 | 3
Headache (Nervous system disorders) | 20 | 16 | 21 | 25 | 38 | 3 | 1 | 4
Depression (Psychiatric disorders) | 6 | 1 | 6 | 5 | 9 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 5 | 2 | 4 | 5 | 7 | 0 | 1 | 2
Hypertension (Vascular disorders) | 4 | 5 | 5 | 2 | 7 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 6 | 7 | 1 | 12 | 17 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Erythema infectiosum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infected insect bite (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Red blood cell burr cells present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abscess Limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Acute Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anisocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Potassium Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Urea Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Urine Present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breath Sounds Abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bundle Branch Block Left (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervical Dysplasia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eosinophil Count Decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophil Count Increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Excoriation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial Pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemicephalalgia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection Site Erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection Site Extravasation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection Site Inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection Site Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Local Swelling (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower Respiratory Tract Infection (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Macrocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Monocyte Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral Candidiasis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Poikilocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Protein Urine Present (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Red Blood Cell Abnormality (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Red Blood Cell Morphology Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal Tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Smear Cervix Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tension Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thyroid Function Test Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo Positional (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other